CLINICAL TRIAL: NCT06444633
Title: The Impact of Pre-emptive Home Delivery of ORS + Zinc on Treatment for Child Diarrhea: a Cluster Randomized Controlled Trial in Bauchi, Nigeria
Brief Title: The Impact of Pre-emptive Home Delivery of ORS + Zinc on Treatment for Child Diarrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Clinton Health Access Initiative, Nigeria (Other); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HCAAD201
Record Dates: First submitted 2024-05-24; First posted 2024-06-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Diarrhea Toddler
Keywords: Oral Rehydration Salts; Child Diarrhea; Zinc

STUDY DESIGN:
Intervention Model Description: The study is a parallel, cluster randomized controlled trial, randomizing administrative wards in Bauchi, Nigeria to treatment (receiving pre-emptive, free ORS+Zinc co-packs (2 nos) per child under 5 to households, along with information about proper use of ORS and Zinc for treating child diarrhea) or delayed-start control (receiving intervention after the end of the study period).
Who Masked: Outcomes Assessor
Masking Description: The enumerator and the outcomes assessor will be masked to the assignment of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed-start control (No Intervention): Wards randomly assigned to this arm will not receive any intervention until after endline data collection in completed. During the study period, the caregivers in this group will have standard access to ORS and zinc at local health facilities and pharmacies. Some community health workers in control villages could make household visits; however, any delivery of ORS or zinc in the control group is not expected as community health workers are generally not the source of diarrhea treatment.
- Community Sensitization + Household visit + Information + Free pre-emptive distribution of ORS+Zinc (Experimental): Wards randomized to this arm will primarily receive four intervention components as described under the "Intervention" section
  Interventions: Behavioral: Community Sensitization + Household visit + Information + Free pre-emptive distribution of ORS+Zinc

INTERVENTIONS:
Behavioral: Community Sensitization + Household visit + Information + Free pre-emptive distribution of ORS+Zinc — The intervention will involve the following: 1) The communities will be sensitized on the importance of ORS and Zinc use for the treatment of child diarrhea, by the Clinton Health Access Initiative (CHAI). 2) Campaigners recruited by CHAI will visit each household in their catchment area that contain at child under 5 years old. 3) During the distribution visits, the campaigners will train caregivers on the dangers of diarrhea and the importance of ORS and zinc use, among other things (including how to prepare, use, and store ORS/zinc, benefits of the treatments, recommended health behaviors such as seeking care, and encouraging basic handwashing and hygiene practices). The caregivers will also receive a flyer describing the same information in their local language, for future reference. 4) Campaigners will then distribute two ORS and zinc co-packs (each co-pack contains two sachets of ORS and 10 tablets of zinc) for free for each child under the age of five in the household.
  Arms: Community Sensitization + Household visit + Information + Free pre-emptive distribution of ORS+Zinc

SUMMARY:
The aim of this clustered randomized controlled trial is to evaluate whether free and pre-emptive distribution of Oral Rehydration Salts (ORS) and Zinc at home increases the use of ORS to treat diarrhea cases among children under the age of 5 in Bauchi, Nigeria. The primary research questions for the study are:

* RQ1a: Does pre-emptive home delivery with free distribution of ORS and zinc coupled with information about the importance of proper treatment (henceforth referred to as "the intervention") result in greater use of ORS to treat child diarrhea (for children under the age of 5) over the 6 months following the deliveries, relative to the status quo (i.e., in the absence of such an intervention)?
* RQ1b: Does the intervention result in greater use of ORS to treat child diarrhea (for children under the age of 5) over the 12 months following the deliveries, relative to the status quo?
* RQ1.1: How much does the effect of the intervention on use of ORS to treat child diarrhea (for children under the age of 5) change over time?

All wards in Bauchi state will be randomly assigned to one of two groups:

* treatment, where all households with at least one child under the age of 5 will receive free pre-emptive ORS and zinc co-packs - with two ORS sachets and 10 zinc tablets per child - coupled with information about the importance of proper treatment
* delayed-start control, with care as usual during the evaluation period and intervention delivery post evaluation) groups.

A total of 1,732 enumeration areas (EAs) will be sampled across all wards for the study period. Within each EA, 20 eligible households will be randomly sampled for surveys during each wave of data collection: baseline, endline wave 1 (over 1-6 months post intervention), and endline wave 2 (over 7-12 months post intervention). The primary outcomes for the study include the use of ORS to treat child diarrhea over 6 months post-intervention, over 12 months post-intervention, and over each month until 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 15 years old
* Has at least one child under 5 at baseline
* Proficiency in English or Hausa

Exclusion Criteria:

* Living in a temporary home (nomadic population)
* Does not speak English or Hausa
* Unable to give informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103920 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
ORS Use (cases in last 4 weeks) | 1-6 months post intervention
  Self-reported ORS use for a case of child diarrhea that occurred within the last 4 weeks.
ORS Use (cases in last 4 weeks) | 1-12 months post intervention
  Self-reported ORS use for a case of child diarrhea that occurred within the last 4 weeks.
ORS Use (cases in last 4 weeks) | Each month from 1-12 months post intervention
  Self-reported ORS use for a case of child diarrhea that occurred within the last 4 weeks.

SECONDARY OUTCOMES:
Zinc + ORS use | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported Zinc + ORS use for a case of child diarrhea that occurred within the last 4 weeks.
Antibiotic use | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported antibiotic use for a case of child diarrhea that occurred within the last 4 weeks.
Zinc use alone | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported Zinc use for a case of child diarrhea that occurred within the last 4 weeks.
Time to ORS initiation | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Binary and count variables; binary coded to 1 if caregiver started treatment on the same day the diarrhea began; count variable truncated to 7 days.
Exposure to unsafe drinking water | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported use of untreated water to prepare ORS for treating diarrhea experienced by a child who is exclusively breastfed.
Willingness to purchase new ORS packets | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported use of ORS, seeking care, and purchase of ORS among households that experienced at least twice as many diarrhea cases as the number of children under 5.
Child mortality; all cause and from diarrhea | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported mortality (all cause and diarrhea) of children under 5 since intervention
Hospitalization from diarrhea | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Self-reported hospitalization (all cause and diarrhea) of children under 5 since intervention
Number of diarrhea episodes | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Count of episodes of diarrhea experienced by children who had at least one case of diarrhea since intervention.
Care seeking outside the home | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Binary indicator, coded to 1 if caregiver sought care from each type of provider.
Wastage of ORS and zinc packets | 1-6 months post intervention, 1-12 months post intervention, and each month from 1-12 months post intervention
  Binary indicator, coded to 1 for each type of wastage (co-packs being lost, co-packs being stolen, co-packs used for non-diarrhea reasons, co-packs given away)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Wagner, Ph.D., Principal Investigator — RAND; Stephanie Bonds, Ph.D., Principal Investigator — RAND
Locations (1):
- Clinton Health Access Initiative, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a public repository at the end of the study.
Supporting Information: Study Protocol
Time Frame: Indefinitely
Access Criteria: Re-identification of study participants will not be permitted. Other criteria as set by the repository.